CLINICAL TRIAL: NCT00111657
Title: A Phase II Multidose Study of Intravenous PEG-uricase in Patients With Refractory Gout
Brief Title: Pegylated Recombinant Mammalian Uricase (PEG-uricase) as Treatment for Refractory Gout
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John Sundy (Other)
Collaborators: Savient Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, John Sundy, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00006845; FD-R-0002537 (Other: FDA OOPD)
Record Dates: First submitted 2005-05-24; First posted 2005-05-25 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-09

CONDITIONS: Gout
Keywords: Gout; Tophi; Tophaceous gout; Allergy to allopurinol; Post-transplant gout
MeSH Terms: conditions — Gout | interventions — Pegloticase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pegloticase (Experimental): All study participants received intravenous pegloticase at dose of 8 mg, administered every 21 days for a maximum of 5 doses.
  There was no control group for this open label study.
  Interventions: Biological: Pegloticase

INTERVENTIONS:
Biological: Pegloticase — 8 mg of Pegloticase administered IV every 3 weeks; total number of infusions is 5
  Other Names: PEG-uricase; PEGylated recombinant mammalian urate oxidase

SUMMARY:
The purpose of this study is to determine whether PEG-uricase (a chemically modified recombinant mammalian enzyme that degrades uric acid) is effective in controlling hyperuricemia in patients with chronic gout, who cannot tolerate, or have not responded adequately, to conventional therapy for gout.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
Inflammatory arthritis in patients with gout is caused by crystals of monosodium urate (MSU) that form as a result of chronically elevated levels of uric acid in plasma and extracellular fluids. Recurrent attacks can usually be prevented by treatment with drugs that block urate synthesis by inhibiting xanthine oxidase, or that promote uric acid excretion. If for various reasons (noncompliance, drug intolerance, inadequate dosage, or inefficacy) therapy fails to maintain serum urate concentration below about 6 mg/dL, gout can progress to a chronic stage characterized by destructive arthropathy, deposition of urate crystals in soft tissues (tophi), and nephropathy. The management of chronic gout in such patients is often complicated by co-morbidities such as hypertension, heart disease, diabetes, and renal insufficiency, which may limit the use of anti-inflammatory agents to treat arthritis.

Urate levels are low and gout does not occur in species that express the enzyme urate oxidase (uricase), which converts urate to the more soluble and easily excreted compound allantoin. Humans do not express this enzyme owing to a mutation of the uricase gene during evolution. Parenteral uricase is thus a potential means of controlling hyperuricemia and depleting urate stores in patients with chronic, refractory gout. Infusion of recombinant fungal uricase is effective in preventing acute uric acid nephropathy due to tumor lysis in patients with malignancies. However, the short circulating life and potential immunogenicity of fungal uricase prevents its chronic use for treating gout.

PEG-uricase is a recombinant porcine urate oxidase to which multiple strands of polyethylene glycol (PEG) of average molecular weight 10,000 have been attached. "PEGylation" is intended to reduce the immunogenicity of uricase, and greatly prolong its circulating life. This "mammalian" PEG-uricase was non-immunogenic and effective in preventing uric acid nephropathy in a uricase-deficient strain of mice (Kelly et al, J Am Soc Nephrol 12:1001-09, 2001). It has been licensed to Savient Pharmaceuticals for clinical development, and has received Orphan Drug designation for the treatment of refractory gout by the FDA Office of Orphan Product Development.

In a Phase I trial sponsored by Savient Pharmaceuticals in 24 subjects with symptomatic gout, single intravenous (IV) infusions of 0.5 to 12 mg of PEG-uricase were well tolerated, and at doses of 4 mg to 12 mg, were effective in normalizing plasma and urinary uric acid levels over a 21-day period post-infusion. Some subjects in this trial developed antibodies to PEG-uricase, but the only serious adverse events observed were attacks of gout. The present Phase II clinical trial in subjects with refractory gout will evaluate the efficacy, safety, and immunogenicity of PEG-uricase when administered at a dose of 8 mg by IV infusion once every 3 weeks, for a total of 5 infusions. The primary measure of efficacy will be a reduction in plasma uric acid to less than 6 mg/dL, and reduction in the ratio of uric acid to creatinine in urine to <0.2. In addition, the ability of PEG-uricase to lower the total uric acid pool size will be evaluated in a subset of treatment subjects. Uric acid pool size will be measured by a method that involves an infusion of uric acid labeled with N15, a stable (non-radioactive) isotope of nitrogen.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Symptomatic gout
* Serum uric acid >7 mg/dL
* Intolerance of, or inadequate response to, conventional therapy for gout
* Women of childbearing potential must have a negative serum pregnancy test and must use an approved birth control method

Exclusion Criteria:

* End stage renal failure that requires dialysis
* Concurrent use of uric-acid lowering agents
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* A history of anaphylactic reaction to a recombinant protein
* Concurrent use of immunosuppressive therapy (except as needed for prevention of rejection of a transplanted organ, or prednisone at 10 mg a day or less for treatment of gout flares)
* A medical or psychological condition which, in the opinion of the investigator, might create undue risk to the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John S. Sundy, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Kelly SJ, Delnomdedieu M, Oliverio MI, Williams LD, Saifer MGP, Sherman MR, Coffman TM, Johnson GA, Hershfield MS. Diabetes insipidus in uricase-deficient mice: a model for evaluating therapy with poly(ethylene glycol)-modified uricase. J Am Soc Nephrol. 2001 May;12(5):1001-1009. doi: 10.1681/ASN.V1251001. PMID 11316859
- [Background] Sundy JS, Ganson N, Kelly SJ, Scarlett EL, Hershfield MS. A Phase I Study of PEGylated Uricase (Puricase®) in Subjects with Gout. Arthritis Rheum 50(9):S337-S338. 2004
- [Background] Ganson NJ, Kelly SJ, Scarlett E, Sundy JS, Hershfield MS. Control of hyperuricemia in subjects with refractory gout, and induction of antibody against poly(ethylene glycol) (PEG), in a phase I trial of subcutaneous PEGylated urate oxidase. Arthritis Res Ther. 2006;8(1):R12. doi: 10.1186/ar1861. PMID 16356199
- [Result] Hershfield MS, Roberts LJ 2nd, Ganson NJ, Kelly SJ, Santisteban I, Scarlett E, Jaggers D, Sundy JS. Treating gout with pegloticase, a PEGylated urate oxidase, provides insight into the importance of uric acid as an antioxidant in vivo. Proc Natl Acad Sci U S A. 2010 Aug 10;107(32):14351-6. doi: 10.1073/pnas.1001072107. Epub 2010 Jul 26. PMID 20660758
- [Derived] Hershfield MS, Ganson NJ, Kelly SJ, Scarlett EL, Jaggers DA, Sundy JS. Induced and pre-existing anti-polyethylene glycol antibody in a trial of every 3-week dosing of pegloticase for refractory gout, including in organ transplant recipients. Arthritis Res Ther. 2014 Mar 7;16(2):R63. doi: 10.1186/ar4500. PMID 24602182

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm - Pegloticase
Started | 37 (37 consented. 30 initiated treatment. 29 completed at least 1 dose.)
Completed | 21 (Completed all intended doses.)
Not Completed | 16

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm - Pegloticase
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 37
Baseline urate concentration (pUA) [Mean (Standard Deviation); unit: mg/dL] | 10.8 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Plasma Uric Acid to Less Than 6 mg/dL.
Time Frame: Baseline to Day 105
Measure: Number; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 30
Participants | 17

2. Secondary Outcome: Clinical Response: Number of Swollen and Tender Joints
Description: Count of tenderness and swelling of 68 joints
Time Frame: Basline and day 134
Population: 30 subject assesed at baseline. 21 subjects who completed study were assesed at day 134
Measure: Median (Inter-Quartile Range); unit: joints
Groups:
- Pegloticase: All study participants received intravenous pegloticase at dose of 8 mg, administered every 21 days for a maximum of 5 doses.
  There was no control group for this open label study.
  Pegloticase: 8 mg of Pegloticase administered IV every 3 weeks; total number of infusions is 5
Arm/Group | Pegloticase
Number analyzed (Participants) | 30
joints
  Number of Tender joints at baseline | 13 [6 to 21]
  Number of Tender joints at day 134 | 2 [1 to 9]
  Number of Swollen jonts at baseline | 9 [5 to 20]
  Number of Swollen jonts at day 134 | 6 [2 to 11]

3. Secondary Outcome: In a Subset of Subjects Who Volunteer Separately, Change in Uric Acid Pool Size Will be Assessed by a Method That Involves Infusion of Uric Acid Labeled With N15, a Stable (Nonradioactive) Isotope of Nitrogen.
Time Frame: baseline and 7 weeks after last infusion
Population: Data was not collected for this outcome as a result of a separate pilot study demonstrating that the measure was not useful.
Arm/Group | Pegloticase
Number analyzed (Participants) | 0

4. Secondary Outcome: Reduction of the Ratio of Uric Acid:Creatinine in Urine
Time Frame: baseline then weekly
Population: These data were not calculated because the effect size of serum irate reduction in plasma was so robust that there was no utility in this assessment.
Arm/Group | Pegloticase
Number analyzed (Participants) | 0

5. Secondary Outcome: Development of Antibodies to PEG-uricase
Description: Number of patients who developed antibodies to PEG-uricase
Time Frame: baseline, then prior to infusions and 7 wks after last infusion
Population: One subject withdrew prior to completing the first infusion and is not included in this analysis.
Measure: Number; unit: participants
Arm/Group | Pegloticase
Number analyzed (Participants) | 29
participants | 15

6. Secondary Outcome: Infusion 1: Maximum Concentration (Cmax) Value
Description: The highest drug concentration in the blood after the first infusion of study drug.
Time Frame: 2 hours
Population: One subject withdrew prior to completing the first infusion and is not included in this analysis.
Measure: Mean (Standard Deviation); unit: mU/mL
Arm/Group | Single Arm - Pegloticase
Number analyzed (Participants) | 29
mU/mL | 25.6 (5.0)

7. Secondary Outcome: Infusion 1: Minimum Concentration (Cmin)
Description: The lowest drug concentration in the blood after the first infusion of study drug.
Time Frame: 21 days after the infusion
Population: One subject withdrew prior to completing the first infusion and is not included in this analysis.
Measure: Mean (Standard Deviation); unit: mU/mL
Arm/Group | Single Arm - Pegloticase
Number analyzed (Participants) | 29
mU/mL | 4.9 (4.6)

ADVERSE EVENTS:
Time Frame: Day 134
Arm/Group | Single Arm - Pegloticase
Serious Adverse Events (participants affected / at risk) | 4/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm - Pegloticase (N=30)
Gastrointestinal bleeding. (Gastrointestinal disorders) | 1 (1)
Bowel perforation. (Gastrointestinal disorders) | 1 (1)
Death (Cardiac disorders) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm - Pegloticase (N=30)
Hypertension (Cardiac disorders) | 4 (4)
Hypotension (Cardiac disorders) | 2 (2)
Abdominal cramping (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 5 (6)
Indigestion (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 2 (3)
Fever (General disorders) | 2 (3)
Lightheadedness (General disorders) | 1 (2)
Urinary hesitancy (Renal and urinary disorders) | 1 (2)
Toothache (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3)
Infected tophus (Infections and infestations) | 1 (1)
Rectal abscess (Infections and infestations) | 1 (1)
Skin abscess (Infections and infestations) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Tooth abscess (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hyperkalemia (Endocrine disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Charcot joint (Musculoskeletal and connective tissue disorders) | 1 (1)
Draining tophus (Musculoskeletal and connective tissue disorders) | 2 (2)
Gout flare (Musculoskeletal and connective tissue disorders) | 27 (119)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in limb (Musculoskeletal and connective tissue disorders) | 2 (3)
Headache (Nervous system disorders) | 3 (3)
Parasthesia (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Conjunctival injection (Eye disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Decreased libido (Psychiatric disorders) | 1 (1)
Excessive sleepiness (Psychiatric disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Labile affect (Psychiatric disorders) | 2 (2)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest tightness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstructive sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 4 (5)
Foot ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Hair loss (Skin and subcutaneous tissue disorders) | 1 (1)
Leg ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (7)
Swellng of toes (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (3)
Nevi (Skin and subcutaneous tissue disorders) | 1 (1)
Seborrheic keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Edema (Cardiac disorders) | 3 (3)
Hyperglycemia (Endocrine disorders) | 1 (1)
Syncope (Cardiac disorders) | 1 (1)
Chronic gouty arthritis (Musculoskeletal and connective tissue disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No